CLINICAL TRIAL: NCT04967404
Title: The Effect of Phosphatidylserine on Time Trial Performance in Trained Male Cyclists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mark Glaister (Other)
Responsible Party: Sponsor-Investigator, Mark Glaister, Principal Investigator, St Mary's University College
Organization: St Mary's University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: StMarysUC
Record Dates: First submitted 2021-06-11; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: The Focus of the Study is to Investigate the Effects of Phosphatidylserine Supplementation on Exercise Physiology and Cycling Time-trial Performance
MeSH Terms: interventions — Phosphatidylserines

STUDY DESIGN:
Intervention Model Description: Participants matched on cycling time-trial performance and then randomly assigned to treatment or placebo groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experiment will follow a double-blind design where all participants and investigators will be blinded to the treatments given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phosphatidylserine, 800 mg per day, 10 days (Experimental)
  Interventions: Dietary Supplement: Phosphatidylserine
- Maltodextrin, 800 mg per day, 10 days (Placebo Comparator)
  Interventions: Dietary Supplement: Phosphatidylserine

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine — 800 mg per day for 10 days

SUMMARY:
Phosphatidylserine is a phospholipid found in high concentrations in the brain and nervous tissues along with naturally occurring in many foods. It has been extensively studied for its effects on improving cognitive function, learning, memory and alleviating stress. However, more recently it has been proposed that phosphatidylserine could improve exercise capacity. The mechanisms of proposed action are difficult to distinguish because of the limited research and therefore the purpose of this study is to identify the proposed mechanism of action of phosphatidylserine supplementation and to establish whether these mechanisms will have an effect on time trial performance in trained male cyclists.

ELIGIBILITY:
Inclusion Criteria:

* Cyclists
* Maximum oxygen uptake of at least 55 mL/kg/min

Exclusion Criteria:

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants must be trained male cyclists
Enrollment: 20 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-22 (Estimated); Study Completion 2021-09-22 (Estimated)

PRIMARY OUTCOMES:
30 minute cycling time-trial power output on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Mean power output

SECONDARY OUTCOMES:
Oxygen consumption at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using an online breath-by-breath gas analyser
Respiratory exchange ratio at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using an online breath-by-breath gas analyser
Breathing frequency at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using an online breath-by-breath gas analyser
Minute ventilation at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using an online breath-by-breath gas analyser
Blood lactate concentration at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Obtained via capillary puncture and analysed using an automated analyser
Blood glucose concentration at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Obtained via capillary puncture and analysed using an automated analyser
Rating of perceived exertion at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using a 15-point (6-20) scale
Heart rate at four different exercise intensities (40, 50, 60 and 70% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer | From baseline to 11 days post supplementation
  Evaluated using a heart rate monitor

IPD SHARING:
Plan to Share IPD: No